CLINICAL TRIAL: NCT00867347
Title: Randomised Trial of Selective Bladder Preservation Against Radical Excision (Cystectomy) in Muscle Invasive T2/T3 Transitional Cell Carcinoma of the Bladder - Feasibility Study
Brief Title: Radiation Therapy or Surgery in Treating Patients Receiving Chemotherapy for Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000633526; ICR-SPARE; ISRCTN61126465; EU-20907; ICR-CTSU/2006/10002
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage II bladder cancer; stage III bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Active Comparator): Patients undergo a radical cystectomy, including pelvic lymphadenectomy,
  between 4 and 6 weeks after initiating course 4 of chemotherapy.
  Interventions: Procedure: therapeutic conventional surgery
- Arm II (Experimental): Patients with no visible residual tumor (cT0 or pT0) or residual but superficial tumor (pTa, pT1) undergo radiotherapy beginning within 4-6 weeks of day 1 of course 4 and continuing for 6.5 weeks.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Patients undergo radical cystectomy
  Arms: Arm I
Radiation: radiation therapy — Patients undergo radiotherapy
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether radiation therapy is more effective than surgery in treating patients with bladder cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared with surgery in treating patients with bladder cancer who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility and patient acceptability of radical cystectomy vs selective bladder preservation (SBP) after neoadjuvant chemotherapy in patients with muscle-invasive transitional cell carcinoma of the bladder.
* To determine compliance rates of patients with their assigned treatments.
* To determine if bladder preservation is equivalent to radical cystectomy, in terms of overall survival, in responders to neoadjuvant chemotherapy.

Secondary

* To compare the overall survival of patients receiving SBP vs radical cystectomy.
* To determine the rate of salvage cystectomy in patients undergoing bladder preservation.
* To determine and compare the toxicity of treatment in both arms.
* To determine and compare quality of life of patients treated with these regimens.
* To compare locoregional progression-free and metastasis-free survival of patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to cancer center and randomized to 1 of 2 treatment arms. Patients are assessed after completion of 3 courses of pre-study neoadjuvant chemotherapy. Patients with poor response (≥ pT2, residual pT2, macroscopic invasive tumor) undergo immediate radical cystectomy (within 6 weeks fo completing chemotherapy). Patients* with responsive disease (≤ pT1 tumor or macroscopically normal bladder) proceed to course 4 of chemotherapy (on-study) followed by treatment according to randomization arm.

NOTE: *Patients with a clear bladder or those who are unsure of their histological results prior to course 4 also proceed to chemotherapy.

* Course 4 of neoadjuvant chemotherapy: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and cisplatin IV over 4 hours on day 1.
* Arm I (radical cystectomy): Patients undergo a radical cystectomy, including pelvic lymphadenectomy, between 4 and 6 weeks after initiating course 4 of chemotherapy.
* Arm II (selective bladder preservation): Patients with no visible residual tumor (cT0 or pT0) or residual but superficial tumor (pTa, pT1) undergo radiotherapy beginning within 4-6 weeks of day 1 of course 4 and continuing for 6.5 weeks.

Health-related quality of life is assessed periodically.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma (TCC) of the bladder

  * Clinical stage T2-T3, N0, M0
* No widespread carcinoma in situ (CIS) or CIS remote from muscle invasive tumor
* No adenocarcinoma, squamous cell carcinoma (SCC), small cell carcinoma, or other variant histology

  * N.B. squamoid differentiation or mixed TCC/SCC allowed
* No simultaneous upper tract, urethral, or prostatic urethral TCC

  * Direct prostatic urethral extension from bladder primary allowed if not involving prostatic stroma
* Currently receiving 3 courses of gemcitabine hydrochloride-cisplatin or other protocol approved neoadjuvant chemotherapy regimen AND willing and fit to receive a 4th course according to study protocol

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin > 10 g/dL
* WBC > 3,000/mm³
* Platelet count > 150,000/mm³
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST < 1.5 times ULN
* Alkaline phosphatase < 1.5 times ULN
* Not pregnant
* Fit for radical cystectomy or radical radiotherapy
* No prior malignancy within the past 5 years except superficial TCC or CIS
* No untreated hydronephrosis

  * Patients with hydronephrosis are eligible if the kidney/ureter has been stented or nephrostomy has been inserted and renal function has been maintained
* No contraindication to radical radiotherapy (e.g., inflammatory bowel disease, radiosensitivity syndrome, or severe diverticular disease)
* No bilateral total hip replacements
* No significant comorbid medical conditions that would interfere with administration of any protocol treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior pelvic radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of patients randomized over 3 years
Proportion of patients undergoing selective bladder preservation
Proportion of patients undergoing radical cystectomy
Overall survival

SECONDARY OUTCOMES:
Compliance with randomized treatment
Rate of salvage cystectomy after selective bladder preservation
Toxicity as assessed by NCI CTCAE v3.0
Quality of life as assessed by the QLQ-C30 v3.0 questionnaire
Locoregional progression-free, metastasis-free, and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Huddart, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Institute of Cancer Research - Sutton, Sutton, England, United Kingdom

REFERENCES:
- [Result] Paramasivan S, Huddart R, Hall E, Lewis R, Birtle A, Donovan JL. Key issues in recruitment to randomised controlled trials with very different interventions: a qualitative investigation of recruitment to the SPARE trial (CRUK/07/011). Trials. 2011 Mar 15;12:78. doi: 10.1186/1745-6215-12-78. PMID 21406089
- [Result] Huddart RA, Birtle A, Maynard L, Beresford M, Blazeby J, Donovan J, Kelly JD, Kirkbank T, McLaren DB, Mead G, Moynihan C, Persad R, Scrase C, Lewis R, Hall E. Clinical and patient-reported outcomes of SPARE - a randomised feasibility study of selective bladder preservation versus radical cystectomy. BJU Int. 2017 Nov;120(5):639-650. doi: 10.1111/bju.13900. Epub 2017 May 29. PMID 28453896